CLINICAL TRIAL: NCT03514212
Title: Testing an Intervention to Increase Physical Activity in Schizophrenia: A Feasibility and Acceptability Study.
Brief Title: Promoting Physical Activity in People With Schizophrenia.
Acronym: ProActiveS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015/0383; 185550 (Other: IRAS Project ID); DTF/12/12 (Other Grant/Funding Number: Chief Scientist Office); 15-SS-0192 (Other: NHS Lothian REC)
Record Dates: First submitted 2018-03-27; First posted 2018-05-02 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Schizophrenia
Keywords: physical activity; intervention; walking
MeSH Terms: conditions — Schizophrenia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ProActiveS (Experimental): As this was a feasibility study, all participants received the intervention.
  Interventions: Behavioral: ProActiveS

INTERVENTIONS:
Behavioral: ProActiveS — A 12-week behaviour change intervention, during which time participants met with the researcher weekly and used a pedometer to measure step count and completed an activity diary to monitor progress, set goals and plan how to cope with identified barriers.

SUMMARY:
People with schizophrenia die approximately 20 years earlier than those in the general population, and this is mostly due to cardiovascular disease (CVD) and related poor physical health. The risk factors for CVD are significantly more prevalent in people with schizophrenia, but they are largely preventable by, for example, engaging in regular PA. Existing interventions to increase PA in schizophrenia are generally atheoretical and lack manualisation and appropriate evaluation, thus reducing their usefulness to clinical practice.

Drawing on the MRC Guidelines for the development and evaluation of complex interventions, a 12-week intervention was developed and informed by a systematic review of the factors that influence PA in people with schizophrenia and a qualitative study exploring the barriers and motivators to PA (n=10). The feasibility and acceptability of the intervention was then investigated in an uncontrolled pilot study (n=20).

The pilot study demonstrated that the intervention was both feasible and acceptable to people with schizophrenia. The retention rate was 90% (n=18), and reasons given for dropout were work commitments and other illness.

Of the 18 who completed the intervention, 17 (94%) increased their weekly step count, 14 (78%) met current public health guidelines of 10,000 steps per day at some point during the 12 weeks, 10 (56%) experienced some weight loss, 12 (67%) took up an additional health promotion opportunity (e.g., improving diet, stopping smoking, joining a gym) and 13 (72%) took up another form of PA in addition to walking (e.g., swimming).

Participants found the intervention enjoyable and thought it should be offered to everyone with schizophrenia. The intervention also proved to be feasible and acceptable to staff who referred patients to take part. Informal feedback from staff confirmed the need for such a service, particularly for those taking anti-psychotic medication, and indicated that, if it was to be implemented more widely, it would be a popular and useful resource.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or related disorder (e.g., schizoaffective disorder, psychosis)
* Living in the community
* Clinically stable for at least 8 weeks prior to intervention enrolment
* Ability to safely walk unaided

Exclusion Criteria:

* Inability to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability of the intervention. | Post intervention (12 weeks).
  Feasibility and acceptability of the intervention was evaluated using mixed-methods to explore recruitment, delivery, reasons for drop-out, participant feedback (positive and negative), and suggestions for improvement. This was quantitatively assessed by recording the number of eligible participants that agreed to participate and the number of participants that enrolled but dropped out. Participants were also asked to complete a feedback form, which contained space for free text, during the last session of the intervention.

SECONDARY OUTCOMES:
Change in weekly step count. | At baseline and at intervention end point (12 weeks).
  Activity was measured objectively using accelerometers.
Change in activity levels. | Throughout the 12-week intervention.
  Participants used their pedometers to measure daily step count and record totals in their activity diaries. Participants also recorded sedentary time in their activity diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Lawrie, MBChB,FRCPsych, Principal Investigator — University of Edinburgh; Gillian E Mead, MBChB,FRCPEd, Principal Investigator — University of Edinburgh

REFERENCES:
- [Background] McNamee L, Mead G, MacGillivray S, Lawrie SM. Schizophrenia, poor physical health and physical activity: evidence-based interventions are required to reduce major health inequalities. Br J Psychiatry. 2013 Sep;203(3):239-41. doi: 10.1192/bjp.bp.112.125070. PMID 24085733